CLINICAL TRIAL: NCT05714735
Title: Assessment of Superficial Cerebral Venous Structures in Brain Swelling in Patients With Subarachnoid Hemorrhage From Anterior Communicating Artery Aneurysmal
Brief Title: SMCV Assessment on Brain Swelling in Patients With SAH From Ruptured Artery Aneurysm
Acronym: SMCV
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: The People Hospital of Baoan Shenzhen (Other)
Responsible Party: Sponsor
Other Study IDs: BAOAN SMCV in SAH
Record Dates: First submitted 2023-01-27; First posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Arterial Aneurysm
Keywords: Brain Swelling,Subarachnoid Hemorrhage,Artery Aneurysmal
MeSH Terms: conditions — Brain Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Whole-brain venography: Cerevbral venography
  Interventions: Radiation: Cerebral Venography

INTERVENTIONS:
Radiation: Cerebral Venography — Cerebral Venography Observation by DSA examinations

SUMMARY:
Superficial cerebral veins findings in assessment of brain swelling in patients with aneurysmal subarachnoid hemorrhage who underwent intravenenous DSA examinations

DETAILED DESCRIPTION:
Superficial cerebral veins findings in assessment of brain swelling in patients with aneurysmal subarachnoid hemorrhage who underwent intravenenous DSA examinations.To explore the relationship between the structure of middle and superficial cerebral veins in cerebral angiography and cerebral edema after ischemia-reperfusion of anterior circulation with large core infarction.

ELIGIBILITY:
Inclusion criteria:

* age 18-70 years;
* Hunt-Hess grade IV-V on admission; single aneurysm in the anterior circulation; interventional embolization of aneurysm is the first choice, and preoperative ventricular puncture drainage and intracranial pressure probe placement.

Exclusion criteria:

* Hunt-Hess grade I-III on admission;
* patients with blood bubble-like aneurysm or accompanying intracranial hematoma who are not suitable for interventional embolization; those who directly choose craniotomy and clipping;
* poor general condition or combined with pregnancy , malignant tumors, etc.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with anterior circulation aneurysmal subarachnoid hemorrhage
Sampling Method: Non-Probability Sample
Enrollment: 198 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-12-07 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Death | One year
  Death
Bleeding events | One year
  Intracerebral Hemorrhage

SECONDARY OUTCOMES:
Brain swelling | One year
  Brain swelling score

CONTACTS AND LOCATIONS:
Overall Officials: qiaoyu huang, M.D, Study Director — The People Hospital of Shenzhen Baoan
Locations (1):
- The People Hospital of Shenzhen Baoan, Shenzhen, Guangdong, China